CLINICAL TRIAL: NCT00432224
Title: Treatment of Actinic Keratoses With Photodynamic Therapy Using Sunlight Versus Red Light
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KF 01-272867
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2007-02-07 (Estimated); Status verified 2007-02

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Photochemotherapy

INTERVENTIONS:
Procedure: photodynamic therapy

SUMMARY:
The objective of the study is to evaluate the use of sunlight instead of red light during photodynamic therapy of actinic keratoses using methyl aminolevulinate

ELIGIBILITY:
Inclusion Criteria:

* symmetric actinic keratoses in scalp or face

Exclusion Criteria:

* porphyria, pregnancy, breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28
Dates: Start 2006-05; Study Completion 2007-02

CONTACTS AND LOCATIONS:
Overall Officials: Hans Christian Wulf, Professor, MD, Study Director — Bispebjerg Hospital; Merete Hædersdal, MD, PhD, Study Chair — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen NV, Denmark